CLINICAL TRIAL: NCT06121518
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial To Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy Versus D064 or D702 Monotherapy in Essential Hypertension Patients
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy Versus D064 or D702 Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A30_17HT2222
Record Dates: First submitted 2023-10-24; First posted 2023-11-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — 2-(3,4-dimethoxyphenyl)-8-(4-hydroxy-3-methoxyphenyl)-6-methyl-2-isopropyl-6-azaoctanitrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): D064 and D702 Combination Therapy
  Interventions: Drug: D064 and D702, QD
- Comparator Group 1 (Active Comparator): D064 Monotherapy
  Interventions: Drug: D064 and Placebo of D702, QD
- Comparator Group 2 (Active Comparator): D702 Monotherapy
  Interventions: Drug: Placebo of D064 and D702, QD

INTERVENTIONS:
Drug: D064 and D702, QD — Experimental Group Subjects assigned to this group are treated with D064, D702
  Other Names: D064 and D702 Combination Therapy
  Arms: Experimental Group
Drug: D064 and Placebo of D702, QD — Comparator Group Subjects assigned to this group are treated with D064, placebo of D702
  Other Names: D064 Monotherapy
  Arms: Comparator Group 1
Drug: Placebo of D064 and D702, QD — Comparator Group Subjects assigned to this group are treated with D702, placebo of D064
  Other Names: D702 Monotherapy
  Arms: Comparator Group 2

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of D064 and D702 Combination Therapy Versus D064 or D702 Monotherapy in Essential Hypertension Patients

DETAILED DESCRIPTION:
This study is a Randomized, Double-blind, Multi-center, Therapeutic confirmatory, Phase 3 Trial To Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy Versus D064 or D702 Monotherapy in Essential Hypertension Patients

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are 19 years old or older.
2. Subjects who are mean blood pressure measured in the arm selected as the reference arm meets the following criteria:

   * Didn't take antihypertensive drug

     * 140 mmHg ≤ MSSBP(mean sitting SBP) < 180 mmHg
   * Taking antihypertensive drug

     * 130 mmHg ≤ MSSBP(mean sitting SBP) < 180 mmHg
3. Subjects who have voluntarily decided to participate in this clinical trial and signed ICF.

Exclusion Criteria:

1. Subjects with a history of secondary hypertension or suspected secondary hypertension
2. Subjects with symptomatic orthostatic hypotension
3. Subjects with type 1 diabetes or diabetes that is not adequately controlled (HbA1c > 9.0%)
4. Subjects with Severe heart failure(NYHA Class 3,4) etc.,
5. Subjects with a history of unstable angina, moderate or malignant retinopathy, etc., within 6 months at the time of screening
6. Subjects with a history of disability to investigational product ADME at the time of screening
7. Subjects with abnormalities in laboratory test results at the time of screening
8. Subjects with hypersensitivity or history of investigational product and similar drugs
9. Subjects who are required to administer a combination of prohibited drugs specified in this plan during the clinical trial participation period
10. Subjects with a history of drug or alcohol abuse or suspected patient within 24 weeks as of the time of screening
11. Subjects who received other investigational product within 4 weeks of screening visit
12. Pregnant women, lactating women, or Subjects who do not agree to use appropriate contraception during the clinical trial period and for two weeks after the end of administration of the last investigational product
13. Subjects who are unable to participate in this clinical trial at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MSSBP(mean sitting SBP(systolic blood pressure)) | 8 weeks
  Compare experimental group with comparator group

CONTACTS AND LOCATIONS:
Overall Officials: Jinho Shin, M.D, Ph.D, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, Seongdong-gu, South Korea